CLINICAL TRIAL: NCT02197390
Title: An Ecological Approach to Addressing Childhood Obesity Issues in Imperial County
Acronym: Our Choice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1U18DP003377-03 (NIH)
Record Dates: First submitted 2014-07-11; First posted 2014-07-22 (Estimated); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Childhood Obesity
Keywords: Childhood obesity; Latino; Hispanic
MeSH Terms: conditions — Pediatric Obesity | interventions — Exercise; Diet, Healthy; Water; Environment; Policy; Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Health Care plus Public Health (Experimental): The Health Care intervention involves the implementation of an obesity care model within a Federally Qualified Health Center (FQHC) and includes a Family Wellness Program delivered by Community Health Workers (CHWs). The Public Health intervention involves working with early care and education centers, schools, community recreation organizations, and restaurants to promote four health behaviors: fruit and vegetable consumption, physical activity, water consumption, and quality sleep.
  Interventions: Behavioral: Family wellness workshops; Behavioral: Obesity chronic care model; Behavioral: Physical activity, healthy eating, water drinking, healthy sleep promotion; Behavioral: Environment, policy, systems changes in clinic setting only; Behavioral: Environment, policy, and systems changes in schools, early child care education & recreation
- Health Care (Experimental): The Health Care intervention involves the implementation of an obesity care model within a Federally Qualified Health Center (FQHC) and includes a Family Wellness Program delivered by Community Health Workers (CHWs).
  Interventions: Behavioral: Family wellness workshops; Behavioral: Obesity chronic care model; Behavioral: Physical activity, healthy eating, water drinking, healthy sleep promotion; Behavioral: Environment, policy, systems changes in clinic setting only
- Public Health (Experimental): The Public Health intervention involves working with early care and education centers, schools, community recreation organizations, and restaurants to promote four health behaviors: fruit and vegetable consumption, physical activity, water consumption, and quality sleep.
  Interventions: Behavioral: Physical activity, healthy eating, water drinking, healthy sleep promotion; Behavioral: Environment, policy, systems changes in clinic setting only
- Control (Experimental): No intervention.
  Interventions: Behavioral: No intervention

INTERVENTIONS:
Behavioral: Family wellness workshops — Nine family wellness workshops and eight family physical activity sessions facilitated by community health workers.
  Arms: Health Care; Health Care plus Public Health
Behavioral: Obesity chronic care model
  Arms: Health Care; Health Care plus Public Health
Behavioral: Physical activity, healthy eating, water drinking, healthy sleep promotion
  Arms: Health Care; Health Care plus Public Health; Public Health
Behavioral: Environment, policy, systems changes in clinic setting only
  Arms: Health Care; Health Care plus Public Health; Public Health
Behavioral: No intervention — No intervention.
  Arms: Control
Behavioral: Environment, policy, and systems changes in schools, early child care education & recreation
  Arms: Health Care plus Public Health

SUMMARY:
Our Choice is one of three CORD (Childhood Obesity Research Demonstration) studies funded by the Centers for Disease Control and Prevention in 2011 to test multi-sector, multi-level approaches to prevent and control childhood obesity. Our Choice is translating evidence-based approaches for modifying behaviors, policies, systems, and environments to promote fruit and vegetable consumption, physical activity, water consumption, and quality sleep. The ultimate goal is to assist Children's Health Insurance Program-eligible children between 2-12 years old attain a healthy weight. In addition to site-specific intervention and evaluation activities, Our Choice is working with the University of Houston Evaluation Center to conduct a cross-site evaluation on a set of shared measures.

DETAILED DESCRIPTION:
Our Choice is a partnership between a university-affiliated research institute, a federally qualified health center, and a county public health department. We used formative research, advisory committee members' recommendations, and previous research to inform the development of the Our Choice project. Our theory-informed multi-sector, multi-level intervention targets improvements in four health behaviors: fruit, vegetable, and water consumption, physical activity, and sleep. Intervention partners include 1200 families, a federally qualified health center (including three clinics), 26 early care and education centers, two elementary school districts (and 20 elementary schools), three community recreation centers, and three restaurants. Intervention components in all sectors target changes in behaviors, policies, systems, and the social and physical environment. Evaluation activities include assessment of the primary outcome, BMI z-score, at baseline, 12- and 18-months post-baseline, and sector evaluations at baseline, 12, and 24-months.

ELIGIBILITY:
Inclusion Criteria:

* If family had school-age child, child must attend one of the designated Our Choice schools located in one of three designated cities.
* If family had preschool-age child, family must reside in one of three designated cities.
* Children ages 2-11 years old
* Maximum two children per household
* Children above the 5th percentile body mass index
* Family agrees to remain in the area throughout the duration of the study
* Participating parent had to understand English or Spanish

Exclusion Criteria:

* Child has any condition that significantly limits eating or physical activity in a way that interventions would be impacted

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1184 (Actual)
Dates: Start 2012-05; Primary Completion 2016-02 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
BMI z-score change in 1184 children, 2-11 years old, assigned to a Health Care plus Public Health intervention, a Health Care intervention only, a Public Health intervention only, or a control condition | 12-month and 18-month post baseline evaluation; December 2015

SECONDARY OUTCOMES:
Child waist circumference | 12-month and 18-month post baseline evaluation; December 2015
Parent waist circumference | 12-month and 18-month post baseline evaluation; December 2015
Parent body mass index | 12-month and 18-month post baseline evaluation; December 2015
  Weight and height
Parent blood pressure | 12-month and 18-month post baseline evaluation; December 2015

OTHER OUTCOMES:
Health clinic health policy adoption | 12-month and 24-month post baseline sector evaluation; October 2015
  Clinic manager interviews
Health clinic implementation of the assessment and treatment of child overweight and obesity guidelines at a specific percentile | 12-month and 24-month post baseline evaluation; October 2015
  Electronic health records (EHR), attendance sheets of trainings attended by health clinic staff, chronic care days in place at each clinic, EHR modifications for assessment and treatment of childhood overweight and obesity, health message posters installed, satisfaction with aspects of the intervention
Body mass index in early care and education centers | Year 1 and Year 2 of intervention; July 2014
  Height and weight measures of children in 23 early child care and education centers.
Body mass index in elementary schools | Year 1 and year 2 of intervention
  Height and weight measures were collected from Kindergarten, 2nd or 3rd, and 5th grade students from 13 elementary schools.

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe X Ayala, PhD, MPH, Principal Investigator — San Diego State University; Leticia Ibarra, MPH, Study Director — Clinicas de Salud del Pueblo, Inc.; Amy Binggeli-Vallarta, DrPH, RD, Study Director — Imperial County Public Health Department
Locations (2):
- United States (2):
  - Our Choice, El Centro, California
  - San Diego State University Research Foundation, San Diego, California

REFERENCES:
- [Background] Chuang E, Ayala GX, Schmied E, Ganter C, Gittelsohn J, Davison KK. Evaluation protocol to assess an integrated framework for the implementation of the Childhood Obesity Research Demonstration project at the California (CA-CORD) and Massachusetts (MA-CORD) sites. Child Obes. 2015 Feb;11(1):48-57. doi: 10.1089/chi.2014.0049. Epub 2014 Nov 25. PMID 25423618
- [Background] Ayala GX, Ibarra L, Binggeli-Vallarta A, Moody J, McKenzie TL, Angulo J, Hoyt H, Chuang E, Ganiats TG, Gahagan S, Ji M, Zive M, Schmied E, Arredondo EM, Elder JP. Our Choice/Nuestra Opcion: the Imperial County, California, Childhood Obesity Research Demonstration study (CA-CORD). Child Obes. 2015 Feb;11(1):37-47. doi: 10.1089/chi.2014.0080. Epub 2015 Jan 13. PMID 25584664
- [Background] Chuang E, Brunner J, Moody J, Ibarra L, Hoyt H, McKenzie TL, Binggeli-Vallarta A, Cervantes G, Finlayson TL, Ayala GX. Factors Affecting Implementation of the California Childhood Obesity Research Demonstration (CA-CORD) Project, 2013. Prev Chronic Dis. 2016 Oct 20;13:E147. doi: 10.5888/pcd13.160238. PMID 27763831
- [Derived] Schmied EA, Madanat H, Chuang E, Moody J, Ibarra L, Cervantes G, Strong D, Boutelle K, Ayala GX. Factors predicting parent engagement in a family-based childhood obesity prevention and control program. BMC Public Health. 2023 Mar 8;23(1):457. doi: 10.1186/s12889-023-15359-7. PMID 36890461
- See also: Click here for more information about the San Diego State University investigators at the Institute for Behavioral & Community Health. — http://www.ibachsd.org